CLINICAL TRIAL: NCT02881944
Title: Effect of Diet on Gulf War Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ashok Tuteja (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ashok Tuteja, Professor Gastroenterology, VA Salt Lake City Health Care System
Organization: VA Salt Lake City Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00087668
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Gulf War Illness; Diet; IBS; FODMAP
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP (modified healthy) Diet (Experimental): Low FODMAP diet for 3 weeks. Veterans will be provided a diet containing foods low in FODMAP.
  Interventions: Behavioral: Low FODMAP Diet
- High FODMAP (typical healthy) Diet (Experimental): High FODMAP diet for 3 weeks. Veterans will be provided a typically healthy diet following US Dietary Guidelines, containing foods high in FODMAPs
  Interventions: Behavioral: High FODMAP Diet

INTERVENTIONS:
Behavioral: Low FODMAP Diet — Diet low in foods containing Fermentable Oligo-, Di-, and Mono-saccharides and Polyols
  Arms: Low FODMAP (modified healthy) Diet
Behavioral: High FODMAP Diet — Typical diet of foods containing Fermentable Oligo-, Di-, and Mono-saccharides and Polyols
  Arms: High FODMAP (typical healthy) Diet

SUMMARY:
Fermentable Oligo-, Di and Mono-saccharides And Polyols (FODMAPs) are carbohydrates that are poorly digested in intestines. The undigested carbohydrates are fermented in the colon by gut bacteria. Fermentation of these carbohydrates can lead to diarrhea, gas and distension of the colon. Low FODMAP diet effect may be mediated by changing the gut bacteria and/or by production of chemicals that influence Veteran's intestines which then result in reduced disease symptoms.

The goal of this study is to compare a low FODMAP (modified healthy) diet to a high FODMAP (typical healthy) diet for effect on Veterans with IBS and symptoms of Gulf War illness.

DETAILED DESCRIPTION:
Study Design This will be a prospective, blinded randomized clinical trial with two parallel groups. There will be 1-week screening period, 3-week diet treatment and, follow-up one month later while Veterans choose their own diet.

Veterans who were deployed and served in Operation Desert Storm and Desert Shield will be recruited to participate.

The two study diets to be provided to the Veterans and compared are:

Low FODMAP (modified healthy) diet:

High FODMAP (typical healthy) diet:

The FODMAP content of this diet will be higher than low FODMAP diet.

All questionnaires will be answered and measurements performed at baseline, end of treatment and at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Gulf War Veterans
* Men and women age 25-90 years
* Gulf War Illness: Veterans will have Rome III criteria for IBS and two or more of the non-intestinal symptom groups (chronic-once a week or more often-fatigue, insomnia, joint pains, general stiffness, and headache, neurological an mood, respirator and skin symptoms)
* Symptoms of > 6 months duration
* No significant findings on physical examination, complete blood count and clinical chemistry panel
* Normal gross appearance of the colonic mucosa (small colon polyps not an exclusion criteria)
* Veterans with psychological disorders will not be excluded but will be identified for sub-group analysis.

Exclusion Criteria:

* Current evidence of any lower gastrointestinal disorder such as celiac disease or inflammatory bowel disease
* Clinically significant chronic disease: HIV, cardiac, pulmonary, hepatic or renal dysfunction
* Presence of Giardia antigen, and Clostridium difficile toxin in stool
* Current history of drug or alcohol abuse
* Investigator perception of patient's inability to comply with study protocol
* Recent change in gastrointestinal medications
* Subject is currently participating in another research protocol. These subjects will be allowed to enroll after a washout period of one month.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported global Bowel Symptom Score | Baseline and 3 Weeks
  Change in bowel symptom score after 3 weeks of treatment with a Low FODMAP diet or High FODMAP diet.

SECONDARY OUTCOMES:
Change in self-reported Irritable Bowel Syndrome Quality of Life (IBS-QOL) score | Baseline and 3 Weeks
  Change in IBS-QOL score after 3 weeks of treatment with a Low FODMAP diet or High FODMAP diet.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok K Tuteja, M.D., Principal Investigator — George E. Wahlen VA Medical Center
Locations (1):
- George E Wahlen VA Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No